CLINICAL TRIAL: NCT02944643
Title: Mindfulness and Support Group to Improve Patient and Caregiver Burden in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor, GI Section, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAJAJ0019
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Mindfulness; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active group (Experimental): Will get the mindfulness and support groups
  Interventions: Other: Mindfulness and Support Groups

INTERVENTIONS:
Other: Mindfulness and Support Groups

SUMMARY:
Chronic liver disease and cirrhosis pose a huge financial burden to the health care system. This includes the cost of medical care, employment, disability-related issues and reduced survival. Specifically, the complication of cirrhosis known as hepatic encephalopathy (HE) especially hinders quality of life, the performance of activities of daily living and the ability to drive a motor vehicle in affected subjects. The hidden burden to family members and caregivers of these subjects, however, has been all but ignored to date. Evaluation of family members and caregivers is essential. The burden of caring for someone with liver disease can result in added cost for health care for family members and caregivers and is typically not recognized. The importance of the burden to families and family members or caregivers resulting from other neurological diseases such as Alzheimer's has been well evaluated and specific strategies to educate and counsel family members and caregivers have been elaborated. This is important because as the findings of this study have emerged, we have found that both Veterans and non-Veterans with cirrhosis and HE have a poor quality of life, worse socio-economic status and place a significantly higher burden on their family members or caregivers than those without HE

DETAILED DESCRIPTION:
The initial intake visit will include an overall assessment of the situation with the subject and family members or caregivers by the study physician and description of the group therapy. If the subjects and family members or caregivers want to continue, they will be asked to visit with the psychologist individually (subject first, then family member or caregiver, then both) in order to confirm their insight into the disease process and assess their readiness and appropriateness for the group therapy.

All concerns regarding confidentiality and details to be discussed during the group therapy sessions will be reiterated to subjects and family members or caregivers individually. They can then choose to participate or not. If they choose not to participate, they will be seen in 1- 3 months to complete the all tests / questionnaires detailed as in the measurements section

Subjects and family members or caregivers agreeing to participate in group therapy will be required to attend four weekly group therapy sessions in order for them to be considered as group therapy recipients. If they choose to terminate the group at any time, they will be free to do so and will be asked to complete all tests / questionnaires detailed as in the measurements section

GROUP INTERVENTION FORMAT:

Group therapy sessions will be conducted on a weekly basis over a four week period. The group therapy sessions will last approximately one hour. The group will not have a rolling admission meaning members will be required to attend all scheduled group sessions.

Measurements used:

* QOL assessment using Sickness Impact Profile (a 136 item questionnaire)
* Sleep assessment using Pittsburgh Sleep Quality Questionnaire (PQSI) and Epworth Sleepiness Scale (ESS)
* Assessment of Depression and Anxiety using the Beck Questionnaires

Structure of the Groups:

Each group will begin with a review of what was learned in the group before and a review of the concrete goals/homework that the participants set from the last group. The group can work together to identify barriers and strategies.

Second portion of the group will focus on acquiring specific skills. These skills include Qigong (gentle movements), body scan, progressive relaxation, and loving-kindness meditation At the conclusion of the session, subjects, family members or caregivers core skills to be targeted as detailed below will be evaluated by the psychologists running the group.

Core Skills to be Targeted:

I. Stress Management II. Dealing with Depression III. Adjusting to Anxiety IV. Family Health and Changes in Roles

ELIGIBILITY:
Patients

Inclusion Criteria:

1. Cirrhosis proven by radiology, endoscopy (esophageal varices present) or biopsy
2. Able to give informed consent as determined by the study staff
3. Have a family member or caregiver who lives with them that is willing to participate

Exclusion Criteria:

1. Unable to give consent
2. Active psychosis
3. Acute suicidal ideation
4. No identified family member or caregiver

Caregivers/Family members:

Inclusion Criteria:

1. Sharing living space with cirrhotic patient for at least 3 years
2. Able and willing to participate in the groups

Exclusion Criteria:

1. Unfamiliar with patient's routines and does not live in the same space
2. Unwilling to consent or participate

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (patients) | 4 weeks

SECONDARY OUTCOMES:
Beck Anxiety Inventory (patients) | 4 weeks
Zarit Burden Interview (caregivers only) | 4 weeks
Sickness Impact Profile (patients) | 4 weeks
Pittsburgh Sleep Quality Index (patients) | 4 weeks
Epworth Sleepiness Scale (patients) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Mcguire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No